CLINICAL TRIAL: NCT01362751
Title: Orthostatic Hypotension in Elderly Nursing Home Residents
Status: Completed | Type: Observational
Sponsor: Medical Research Foundation, The Netherlands (Other)
Responsible Party: Principal Investigator, Kornelis J.J. van Hateren, MD, Medical Research Foundation, The Netherlands
Other Study IDs: OH_TMZ_2010
Record Dates: First submitted 2010-10-07; First posted 2011-05-30 (Estimated); Last update posted 2012-09-05 (Estimated); Status verified 2012-09

CONDITIONS: Orthostatic Hypotension
MeSH Terms: conditions — Hypotension, Orthostatic

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Nursing home residents: In this study, patients from both the somatic and the psychogeriatric department are included. For the primary endpoint 'successful rehabilitation' only the patients from the somatic departments are included.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This study is an observational cohort study > no interventions

SUMMARY:
In this study the investigators aimed

1. to investigate the prevalence of orthostatic hypotension in elderly nursing home residents.
2. to investigate whether the presence of orthostatic hypotension influences the chance of successful rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* nursing home resident

Exclusion Criteria:

* patients at the palliative department
* life expectancy < 4 weeks
* patients only temporarily admitted to the nursing home

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Nursing home residents
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2010-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Orthostatic hypotension | Baseline
  Orthostatic hypotension is defined by consensus as a fall in blood pressure of at least 20 mmHg systolic or 10 mmHg diastolic within 3 minutes in the upright position
Successful rehabilitation | After 5 years
  Successful rehabilitation is defined as whether the patient is able to return to his/her home or another location (but not a nursing home) after discharge from the nursing home. Unsuccessful rehabilitations implies that the patients becomes a long-stay nursing home resident.

SECONDARY OUTCOMES:
All-cause and Cardiovascular mortality | Date of death
Quality of life | Measured at baseline and after 1 year
  Quality of life is measured using the RAND-36 questionnaire.
Fall incidents | After 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Nursing home TriviumMeulenbeltZorg, location Borsthuis, Hengelo, Netherlands

REFERENCES:
- [Derived] Hartog LC, Cizmar-Sweelssen M, Knipscheer A, Groenier KH, Kleefstra N, Bilo HJ, van Hateren KJ. The association between orthostatic hypotension, falling and successful rehabilitation in a nursing home population. Arch Gerontol Geriatr. 2015 Sep-Oct;61(2):190-6. doi: 10.1016/j.archger.2015.05.005. Epub 2015 May 18. PMID 26026216